CLINICAL TRIAL: NCT04736069
Title: The Cost-effectiveness of Inpatient and Outpatient Physical Therapy Programs in Knee Osteoarthritis
Brief Title: Which Physical Therapy Program is Cost-effective in Knee Osteoarthritis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Nihan Cuzdan, Doctor, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UfukUniv
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee
Keywords: cost-effectiveness; knee; osteoarthritis; physical therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Group 1 received 21 sessions of inpatient physical therapy program including electrotherapy, superficial- deep heat applications and basic knee exercise program. Group 2 received the same physical therapy program at outpatient clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient physical therapy program (Active Comparator): The group received 21 sessions of physical therapy program including electrotherapy, superficial- deep heat applications and basic knee exercise program at inpatient clinic.
  Interventions: Other: Physical therapy program
- Outpatient physical therapy program (Active Comparator): The group received the same physical therapy program including electrotherapy, superficial-deep heat applications and basic knee exercise program at outpatient clinic.
  Interventions: Other: Physical therapy program

INTERVENTIONS:
Other: Physical therapy program — In the physical therapy program, 20 minutes of hot pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS; 30 to 40 Hz), 6 minutes of ultrasound (US; 1 MHz, 1 to 1.5 Watt/cm2) therapy were applied to both groups. Both of the programs were supervised by physical therapists. A combined range of motion and strengthening exercises were given to both groups to be performed two times a day.

SUMMARY:
Knee osteoarthritis (OA) is a disease with significant levels of socioeconomic burden to the society. P The non-pharmacologic interventions in knee OA include weight loss, exercise, and physical therapy. In this study, we aimed to to compare the cost-effectiveness of inpatient and outpatient physical therapy programs in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a major problem for society with a heavy economic burden. Especially in the elderly population, integrated rehabilitation programs are frequently used to improve patients' symptoms and quality of life. To estimate the costs and utility of the rehabilitation programs may help clinicians decide optimal treatment strategy with proper usage of resources. Therefore, we aimed to to compare the cost-effectiveness of inpatient and outpatient physical therapy programs in patients with knee osteoarthritis.The study included 52 patients with the diagnose of knee osteoarthritis. Patients were divided into two groups. Group 1 (n=30) received 21 sessions of inpatient physical therapy program including electrotherapy, superficial- deep heat applications and basic knee exercise program. Group 2 (n=22) received the same physical therapy program at outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

-Knee OA diagnosed patients based on American College of Rheumatology Criteria

Exclusion Criteria:

* visual disturbances
* malignancy
* inflammatory rheumatic diseases
* pregnancy
* advanced cardiovascular, kidney or liver pathologies
* uncontrolled hypertension
* patients who had injuries in their lower extremities
* patients who underwent under total hip or knee prosthetic surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2013-01-30 (Actual); Study Completion 2013-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nihan CUZDAN, MD, Principal Investigator — Ufuk University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
The authors will consider providing data for all individual requests after the publication. Requests can be done through e-mail. All individual requests will be evaluated and the data will be shared by the principal investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication
Access Criteria: The authors will consider providing data for all individual requests after the publication.
URL: http://'nihancuzdan@hotmail.com

REFERENCES:
- [Background] Dieppe PA, Lohmander LS. Pathogenesis and management of pain in osteoarthritis. Lancet. 2005 Mar 12-18;365(9463):965-73. doi: 10.1016/S0140-6736(05)71086-2. PMID 15766999
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Hendrich AL, Bender PS, Nyhuis A. Validation of the Hendrich II Fall Risk Model: a large concurrent case/control study of hospitalized patients. Appl Nurs Res. 2003 Feb;16(1):9-21. doi: 10.1053/apnr.2003.YAPNR2. PMID 12624858

RESULTS

PARTICIPANT FLOW:
Groups:
- Inpatient Physical Therapy: Patients who received physical therapy and rehabilitation program at inpatient clinic
- Outpatient Physical Therapy: Patients who received physical therapy and rehabilitation program at outpatient clinic
Period: Overall Study
Arm/Group | Inpatient Physical Therapy | Outpatient Physical Therapy
Started | 30 | 30
Completed | 30 | 22
Not Completed | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Inpatient Physical Therapy: Group 1 received 21 physical therapy sessions, including electrotherapy, superficial-deep heat applications, and a basic knee exercise program at inpatient clinic.
- Outpatient Physical Therapy: Group 2 received 21 physical therapy sessions, including electrotherapy, superficial-deep heat applications, and a basic knee exercise program at outpatient clinic.
- Total: Total of all reporting groups
Arm/Group | Inpatient Physical Therapy | Outpatient Physical Therapy | Total
Number analyzed (Participants) | 30 | 22 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (12.2) | 61.0 (14.1) | 64.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 16 | 43
  Male | 3 | 6 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 30 | 22 | 52
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (4.0) | 26.8 (4.3) | 28.8 (4.5)
Occupation [Count of Participants; unit: Participants]
  unemployed | 29 | 18 | 47
  working | 1 | 4 | 5
Occupational intensity [Count of Participants; unit: Participants]
  light | 28 | 17 | 45
  moderate | 2 | 4 | 6
  heavy | 0 | 1 | 1
Trauma history presence [Count of Participants; unit: Participants]
  present | 6 | 5 | 11
  absent | 24 | 17 | 41
Kellgren Lawrence Grading [Count of Participants; unit: Participants] — Kellgren-Lawrence classification system is used for osteoarthritis grading; grade: 0: none; grade:1 doubtful, grade 2: minimal, grade 3: moderate, grade 4:severe
  Participants
    grade 1/2 | 10 | 14 | 24
    grade 3 | 14 | 5 | 19
    grade 4 | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Pain; Visual Analog Scale (VAS)
Description: Patients were requested to sign their pain level on a 10 cm horizontal line with terminal ends of 'no pain' and 'the worst pain'
Time Frame: Change from Baseline VAS scores at 6 months
Measure: Median (Inter-Quartile Range); unit: cm
Groups:
- Inpatient Physical Therapy: The group received 21 sessions of physical therapy program including electrotherapy, superficial- deep heat applications and basic knee exercise program at inpatient clinic.
  Physical therapy program: In the physical therapy program, 20 minutes of hot pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS; 30 to 40 Hz), 6 minutes of ultrasound (US; 1 MHz, 1 to 1.5 Watt/cm2) therapy were applied to both groups. Both of the programs were supervised by physical therapists. A combined range of motion and strengthening exercises were given to both groups to be performed two times a day.
- Outpatient Physical Therapy: The group received the same physical therapy program including electrotherapy, superficial-deep heat applications and basic knee exercise program at outpatient clinic.
  Physical therapy program: In the physical therapy program, 20 minutes of hot pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS; 30 to 40 Hz), 6 minutes of ultrasound (US; 1 MHz, 1 to 1.5 Watt/cm2) therapy were applied to both groups. Both of the programs were supervised by physical therapists. A combined range of motion and strengthening exercises were given to both groups to be performed two times a day.
Arm/Group | Inpatient Physical Therapy | Outpatient Physical Therapy
Number analyzed (Participants) | 30 | 22
cm | 4 [3 to 6] | 4 [2 to 5]

2. Primary Outcome: Physical Function; Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index
Description: WOMAC questionnaire includes five items for pain, two for stiffness, and 17 for functional limitation (score range 0-68). All the items are scored on a scale of 0-4, with higher scores indicating a higher level of symptoms or physical disability.
Time Frame: Change from Baseline WOMAC scores at 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Inpatient Physical Therapy | Outpatient Physical Therapy
Number analyzed (Participants) | 30 | 22
score on a scale | 26.5 [16 to 38] | 18 [12 to 38]

3. Primary Outcome: Fall Risk Assessment; Hendrich II Fall Risk Scale
Description: The scale includes seven items. These items are confusion & disorientation, depression, change in excretion, dizziness, gender, antiepileptic & benzodiazepine use, and get up and walk test. The final score is the sum of these scores; (the score range is between 0-16; 16 is the highest possible score) Patients five or more scores on the scale are considered to be at high risk.
Time Frame: Change from Baseline Hendrich II Fall Risk Scale at 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Inpatient Physical Therapy | Outpatient Physical Therapy
Number analyzed (Participants) | 30 | 22
score on a scale | 1 [0 to 2] | 1 [0 to 2]

4. Primary Outcome: Quality of Life; Short-Form 36-General Health
Description: Short-Form 36 (SF-36) which is composed of eight multi-item scales as bodily pain, physical functioning, social functioning, role-physical, role-emotional, vitality, general health, mental health. Each score of these scales ranging from 0 to 100; higher scores indicating higher QoL.
Time Frame: Change from Baseline Short-Form 36 scores at 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Inpatient Physical Therapy: The group received 21 sessions of physical therapy program including electrotherapy, superficial- deep heat applications and basic knee exercise program at inpatient clinic.
  Physical therapy program: 20 minutes of hot pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS; 30 to 40 Hz), 6 minutes of ultrasound (US; 1 MHz, 1 to 1.5 Watt/cm2); A combined range of motion and strengthening exercises/two times a day
- Outpatient Physical Therapy: The group received the same physical therapy program including electrotherapy, superficial-deep heat applications and basic knee exercise program at outpatient clinic.
  Physical therapy program: 20 minutes of hot pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS; 30 to 40 Hz), 6 minutes of ultrasound (US; 1 MHz, 1 to 1.5 Watt/cm2); A combined range of motion and strengthening exercises:two times a day.
Arm/Group | Inpatient Physical Therapy | Outpatient Physical Therapy
Number analyzed (Participants) | 30 | 22
score on a scale | -7.5 [-20 to 0] | -7.5 [-20 to 0]

5. Primary Outcome: Median Total Cost Per Participant for Health Care
Description: median total expenses for health care at the end of the study
Time Frame: baseline-six months
Measure: Median (Full Range); unit: euros
Groups:
- Inpatient Physical Therapy: The group received 21 sessions of physical therapy program including electrotherapy, superficial- deep heat applications and basic knee exercise program at inpatient clinic.
  Physical therapy program:, 20 minutes of hot pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS; 30 to 40 Hz), 6 minutes of ultrasound (US; 1 MHz, 1 to 1.5 Watt/cm2) therapy were applied to both groups. A combined range of motion and strengthening exercises; two times a day.
- Outpatient Physical Therapy: The group received the same physical therapy program including electrotherapy, superficial-deep heat applications and basic knee exercise program at outpatient clinic.
  Physical therapy program: 20 minutes of hot pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS; 30 to 40 Hz), 6 minutes of ultrasound (US; 1 MHz, 1 to 1.5 Watt/cm2) therapy were applied to both groups. A combined range of motion and strengthening exercises; two times a day.
Arm/Group | Inpatient Physical Therapy | Outpatient Physical Therapy
Number analyzed (Participants) | 30 | 22
euros | 552.4 [497.2 to 1372.5] | 276.3 [218.0 to 1023.6]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Skin and Subcutaneous Tissue Disorders
Arm/Group | Inpatient Physical Therapy | Outpatient Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Informed Consent Form (2010-10-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT04736069/ICF_000.pdf